CLINICAL TRIAL: NCT03917836
Title: Helicobacter Pylori Eradication Improves Endoscopic Detection Of Dysplasia On Visible Gastric Lesions In Over Middle-Aged Patients
Brief Title: Dysplasia Detection and Helicobacter Pylori Eradication
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Candiolo Cancer Institute - IRCCS (Other)
Responsible Party: Principal Investigator, alba panarese, Principal investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: 67/2018
Record Dates: First submitted 2019-04-13; First posted 2019-04-17 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Precancerous Gastric Lesions; Dysplasia Detection
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Gastric biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: endoscopy and histology — diagnostic evaluation of chronic gastritis

SUMMARY:
The investigators in the present study, aimed to assess the efficacy of both White-Light Endoscopy with High Resolution Endoscopy-Narrow-band imaging in the diagnosis of Premalignant Gastric Conditions, before and after Helicobacter pylori-eradication. A prospective study was performed in our institution involving the regular use of high resolution gastroscopes with and without Narrow-band imaging. From May 2018 to April 2019, all patients that received an endoscopic diagnosis of Helicobacter pylori-related gastritis with/without Premalignant Gastric Conditions by an expert endoscopist, were reassessed by White-Light Endoscopy and High Resolution Endoscopy-Narrow-band imaging, including biopsy samples according to the Sydney system, six months later after the proved Helicobacter pylori-eradication.

DETAILED DESCRIPTION:
Helicobacter pylori infection is commonly responsible for Premalignant Gastric Conditions such as chronic atrophic gastritis and Intestinal Metaplasia, which are strongly associated, when located in antrum and corpus, to the evolution into dysplasia and into the Lauren intestinal-type of Gastric Carcinoma.

Many studies have linked gastric carcinogenesis to genes, genetic variations of the host, as well as to Helicobacter pylori induced inflammation of gastric mucosa. In addition, hostile Helicobacter pylori strains have been considered responsible for more severe degrees of inflammation and more rapid progression to intestinal-type gastric cancer, in genetically predisposed subjects. Nowadays, Premalignant Gastric Conditions detection and surveillance has been considered a cost-effective strategy only in intermediate or high risk regions, for the prevention of high-grade dysplasia and gastric cancer. Anyway, conflicting results deriving from "long-term" endoscopic surveillances (ranging between 2-16 years), have shown that Helicobacter pylori eradication was effective in reducing the prevalence of advanced-Premalignant Gastric Conditions, as well as histological progression of early-Premalignant Gastric Conditions, decreasing gastric cancer incidence. The current European guidelines recommend Helicobacter pylori eradication in at high-risk subjects.

Nevertheless, even after Helicobacter pylori eradication, the risk for Premalignant Gastric Conditions/malignant lesions progresses on long-term follow-up. An adequate upper gastrointestinal endoscopy should include at least four non-targeted biopsies at the lesser and greater curvature, and at the antrum-corpus for Helicobacter pylori infection diagnosis and for the optimal detection/staging of advanced-Premalignant Gastric Conditions, which are randomly distributed throughout the stomach. Additional target biopsies of visible suspected lesions are recommended, since low/high grade dysplasia may appear as endoscopically evident, depressed or raised lesions. Several studies showed that Magnification Chromoendoscopy and Narrow-band imaging with or without magnification could be more accurate than White-Light Endoscopy alone, when performed by expert endoscopists, in diagnosing and differentiating Premalignant Gastric Conditions/lesions, by guiding biopsies for staging atrophic/metaplastic changes and by targeting neoplastic lesions, even if random biopsies may be useful in detecting some cases undetectable by Narrow-band imaging alone, and therefore both White-Light Endoscopy with Narrow-band imaging are suggested. Therefore, as a result of many studies, high definition endoscopy with Chromoendoscopy is considered better than high definition White-Light Endoscopy alone in diagnosing Premalignant Gastric Conditions and early neoplastic lesions, whereas virtual Chromoendoscopy, with or without magnification, should be used for the diagnosis of Premalignant Gastric Conditions. For patients with indefinite diagnosis for dysplasia, or with dysplasia resulted from random biopsies without "apparent" endoscopically visible lesions, the current guidelines suggest a relatively immediate endoscopic reassessment with High Resolution Endoscopy-Narrow-band imaging, to exclude a misdiagnosed low/high grade dysplasia on visible lesion or an early-gastric cancer, differently from the previous guidelines, which advised for the same patients only endoscopic follow-up within 1 year after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* HP-related symptoms
* Gastritis with/without PGC by gastric biopsies and/or by non-invasive tests

Exclusion Criteria:

* Absence of informed consent
* Past gastric cancer or gastric related surgery
* Not being able to perform at least five biopsies during the endoscopic exam
* Relevant comorbidities (such as cardiac, respiratory, chronic renal insufficiency, chronic liver disease, psychiatric conditions, anticoagulant therapy or coagulation disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients that received an endoscopic diagnosis of Helicobacter pylori-related gastritis by an expert endoscopist
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Rate of dysplasia before and after Helicobacter pylori eradication | six months
  diagnostic performance of High Resolution Wight Light Endoscopy with High Resolution Endoscopy Narrow Band Imaging, in detecting Precancerous Gastric Conditions on an interim endoscopic surveillance

SECONDARY OUTCOMES:
The prevalence concordance among the endoscopic (Kimura Takemoto grades, EGGIM scales) and histological findings (OLGA grade, OLGIM grade, dysplasia according WHO classification) | six months
  Concordance among endoscopic and histological findings

CONTACTS AND LOCATIONS:
Locations (1):
- Alba Panarese, Noci, Apulia, Italy

IPD SHARING:
Plan to Share IPD: No